CLINICAL TRIAL: NCT03136224
Title: Comparison of Short and Long Term Complications According to the Circumcision Technique Applied During the Childhood
Brief Title: Examination of Short and Long Term Complications of Thermocautery, Plastic Clamping and Surgical Circumcision Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocatepe University (Other)
Responsible Party: Principal Investigator, Ahmet Ali Tuncer, Asst Prof Dr, Kocatepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2011-KAEK-2. 2016/3:35
Record Dates: First submitted 2017-04-23; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Circumcision, Male
Keywords: circumcision; Thermocautery; Clamp; Surgical Circumcision

STUDY DESIGN:
Intervention Model Description: Thermocautery group Plastic clamping group Classic (Surgical) circumcision group
Who Masked: Outcomes Assessor
Masking Description: Statistician was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thermocautery (Experimental): In the thermocautery method, a digital thermocautery device (Thermo-Med TM 802-B, Thermo Medikal, Adana, Turkey) with 6 different temperature settings was used. Circumcision was performed in the same way as the surgical circumcision. Only cutting and bleeding intervention was done by using a thermocautery device. Cutting was performed by making the appropriate heat adjustment according to the age of the child and the thickness of the glans. Hemorrhage control was performed with a thermocautery device and then the skin-mucosa integrity was ensured by using a 5/0 absorbable suture
  Interventions: Device: Thermocautery
- Plastic Clamping (Active Comparator): Alisklamp (Alisklamp, Abagrup Health Services Ltd, Ankara, Turkey) was used in the plastic clamp technique. The clamp size was chosen according to the diameter of the penis of the patient. The clamp was inserted into the glans and then the skin and the mucosa were pulled to the appropriate size and clamped. The skin and mucosa were excised from the distal part of the clamp with the aid of a lancet. After the operation, the clamp was removed on the 4th day
  Interventions: Device: Plastic Clamping
- Surgical Circumcision (Sham Comparator): In classical surgical circumcision, foreskin was hung up with the clamp. The outer skin and secondly the mucosa was cut by using scissors. Following the hemorrhage intervention, the skin-mucosa integrity was sutured by using the 5/0 absorbable suture. Medical dressing was done.
  Interventions: Device: Surgical Circumcision

INTERVENTIONS:
Device: Thermocautery
  Other Names: Experimental
  Arms: Thermocautery
Device: Plastic Clamping
  Other Names: Active comparator; Alisklamp
  Arms: Plastic Clamping
Device: Surgical Circumcision
  Other Names: sham comparator
  Arms: Surgical Circumcision

SUMMARY:
Since circumcision is a significant workload for surgeons working at the rural state hospitals in Turkey, the use of circumcision techniques that are easy to implement and have low complications is becoming widespread. In this study, thermocautery, plastic clamping, and conventional (open surgical) circumcision techniques were compared to each other in terms of their short and long term complications.

DETAILED DESCRIPTION:
The study was carried out in accordance with the Helsinki declaration rules, with the approval of the local ethics committee. Male patients who applied to Hakkari State Hospital and Yüksekova State Hospital pediatric surgery clinics between May 2014 and May 2015 for the circumcision operation were analyzed retrospectively by using the hospital registry system. Patients were evaluated in terms of age groups, accompanying pathologies, anesthesia techniques, duration of the surgery, complication rates, and circumcision techniques. Data obtained from the study were transferred to a computer environment and assessed with the help of Statistical Package for Social Sciences Version 19.0. Chi-square test was used to evaluate categorical data and Mann-Whitney U test was used to evaluate quantitative variables. The distribution of the data was tested by using one of the normality tests such as Shapiro-Wilk test in case of the comparison of surgical time. Kruskal Wallis test was used for nonparametric tests in group comparisons when data were not normally distributed. The Dunn test was used as a post-hoc test when different groups were determined. P <0.05 was considered statistically significant.

Circumcision was performed by a pediatric surgeon and an assistant health professional under sterile conditions in the operating room or circumcision room.

Penile block and local infiltration anesthesia (penile ring block, penile dorsal nerve block) were performed to all other patients with Bupivacaine, and Prilocaine. Open surgery, thermocautery, and plastic clamp (Alisklamp) methods were used as circumcision techniques.

In classical surgical circumcision, foreskin was hung up with the clamp. The outer skin and secondly the mucosa was cut by using scissors. Following the hemorrhage intervention, the skin-mucosa integrity was ensured by using the 5/0 absorbable suture. Medical dressing was done.

Alisklamp was used in the plastic clamp technique. The clamp size was chosen according to the diameter of the penis of the patient. The clamp was inserted into the glans and then the skin and the mucosa were pulled to the appropriate size and clamped. The skin and mucosa were excised from the distal part of the clamp with the aid of a lancet. After the operation, the clamp was removed on the 4th day.

In the thermocautery method, a digital thermocautery device with 6 different temperature settings was used. Circumcision was performed in the same way as the surgical circumcision. Only cutting and bleeding intervention was done by using a thermocautery device. Cutting was performed by making the appropriate heat adjustment according to the age of the child and the thickness of the glans. Hemorrhage control was performed with a thermocautery device and then the skin-mucosa integrity was ensured by using a 5/0 absorbable suture.

Routine warm sitting pool and daily medical dressing were recommended after circumcision. Furthermore, it was recommended to patients with phimosis to apply epithelium cicatrising cream. On the 10th postoperative day, all patients were recruited for routine control. Patients with complications were followed up for a long term. Complications were treated.

ELIGIBILITY:
Inclusion Criteria:Circumcised by Thermocautery, Alisklamp and surgical circumcision techniques

-

Exclusion Criteria: Other circumcision Techniques (Tara, Mogen clamp...) excluded

Ages: 1 Week to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2062 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | May 2014 and May 2015 (circumcised in 1 year period)
  The diversity in circumcision techniques is because of the search for a more practical, cheaper, safer, and less complicated technique. In this study, complications of circumcisions performed by pediatric surgeon specialists by using three different techniques (thermocautery, alisklamp, and surgical circumcision) in two different hospitals in Turkey were investigated retrospectively.

SECONDARY OUTCOMES:
Surgical processing time | May 2014 and May 2015 (circumcised in 1 year period)
  Surgical processing time of groups were analyzed retrospectively by using the hospital registry system

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Ali Tuncer, Asst Prof Dr, Principal Investigator — Afyon Kocatepe University

IPD SHARING:
Plan to Share IPD: Yes